CLINICAL TRIAL: NCT06014723
Title: Balloon angiopLasty for Intracranial Atherosclerotic Minor Stroke/TIA: a Prospective, Multi-center, Register Study
Brief Title: Balloon angiopLasty for Intracranial Atherosclerotic Minor Stroke/TIA
Status: Recruiting | Type: Observational
Sponsor: Shouchun Wang, MD, PhD (Other)
Collaborators: The General Hospital of Northern Theater Command (Other)
Responsible Party: Sponsor-Investigator, Shouchun Wang, MD, PhD, Chief physician of the Department of Neurology, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: BLAST
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: The observation group received early submaximal balloon angioplasty and medical therapy.
  Interventions: Procedure: Submaximal balloon angioplasty
- Control group: The control group received only medical therapy.

INTERVENTIONS:
Procedure: Submaximal balloon angioplasty — The goal of submaximal balloon angioplasty is to use the balloon to improve the stenosis of the criminal artery by more than 20%.
  Groups: Observation group

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of early submaximal balloon angioplasty combined with medical therapy vs medical therapy alone for minor stroke/transient ischemic attack with intracranial atherosclerosis etiology.

DETAILED DESCRIPTION:
In this study, 416 patients with minor strokes or transient ischemic attacks due to symptomatic intracranial atherosclerotic stenosis within one week of the onset of last ischemic symptoms from 20 centers in China were enrolled. The observation group received early submaximal balloon angioplasty, while the control group received only medical therapy. Two groups will be followed up for 1 year to evaluate the safety and efficacy of early submaximal balloon angioplasty combined with medical therapy vs medical therapy alone for minor stroke / transient ischemic attack with intracranial atherosclerosis etiology.

ELIGIBILITY:
Inclusion Criteria:

1. age range of 30-80 years;
2. symptomatic ICAS (C4-C7 segments of ICA, M1 segment of the MCA, V4 segment of the VA, and BA) with 70%-99% stenosis confirmed by DSA;
3. minor stroke (NIHSS score ≤5) within 1 week of onset or from symptom exacerbation (NIHSS score increased by ≥2 points) or intermediate- to high-risk TIA, defined as ABCD2 score ≥4 within 1 week of the last symptom episode;
4. diameter of the culprit artery ranging from 2.0 to 4.5mm, and the length of the stenosis≤14mm;
5. mRS ≤ 2 before endovascular treatment；
6. no large ischemic region found on CT or MRI (ASPECTS≥ 6 or pc-ASPECTS ≥8)；
7. written informed consent obtained from the patient or legally responsible person.

Exclusion Criteria:

1. allergy to contrast media;
2. non-atherosclerotic disease-related stenosis, such as arterial dissection, Moya-Moya disease, and arteritis;
3. penetrating branch lesion ipsilateral to the target lesion (infarction caused by penetrating branch occlusion is defined as stenosis of the MCA or BA, but only with simple basal ganglia or brainstem/thalamic infarction);
4. presence of severe stenosis of the extracranial segment on the side of the target lesion;
5. previous endovascular treatment of the ipsilateral vessel;
6. presence of intracranial aneurysms, tumors, and vascular malformations;
7. any form of ipsilateral intracranial hemorrhage within 3 months and contralateral intracranial hemorrhage within 2 weeks;
8. presence of atrial fibrillation, severe heart dysfunction, liver or kidney dysfunction; patients with tumors and serious diseases whose expected survival time is ≤ 1 year;
9. hemoglobin ≤ 100g/L, platelet count ≤ 100×10^9/L, INR> 1.5 (irreversible), coagulopathy or irremediable bleeding factors;
10. uncontrollable hypertension: systolic blood pressure >185 mmHg and/or diastolic blood pressure >110 mmHg;
11. poor glycemic control (random blood glucose > 22.2 mmol/L);
12. history of major surgery within 30 days prior to enrollment or surgery plan within 90 days after enrollment;
13. pregnancy or lactation;
14. other conditions that the researchers think make the patient unsuitable for the study.

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with minor stroke/transient ischemic attack.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroke or death within 30 days or ischemic stroke in the culprit artery territory from 30 days to 1 year | 30 days, 1 year
  Stroke or death within 30 days or ischemic stroke in the culprit artery territory from 30 days to 1 year

SECONDARY OUTCOMES:
Stroke or death within 30 days after enrollment | 30 days
  Stroke or death within 30 days after enrollment
Ischemic stroke in the territory of criminal artery from 30 days to 1 year after enrollment | 1 year
  Ischemic stroke in the territory of criminal artery from 30 days to 1 year after enrollment
Restenosis rate of criminal artery within 1 year after enrollment | 1 year
  Restenosis rate of criminal artery within 1 year after enrollment
Evaluation of neurological function improvement within 90 days of enrollment | 90 days
  Evaluation of neurological function improvement within 90 days of enrollment

OTHER OUTCOMES:
Intracranial hemorrhage within 30 days of enrollment | 30 days
  Intracranial hemorrhage within 30 days of enrollment
Complications associated with endovascular therapy | 24 hours, discharge, 30 days, 90 days, and 1 year after enrollment
  Complications associated with endovascular therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Qi S, Liu L, Yue FX, Qiu J, Li W, Li C, Nguyen TN, Wei M, Chen HS, Wang SC. Balloon angiopLasty for intracranial Atherosclerotic minor Stroke/TIA (BLAST): study protocol for a multicenter prospective cohort study. Front Neurol. 2024 May 24;15:1385546. doi: 10.3389/fneur.2024.1385546. eCollection 2024. PMID 38854963